CLINICAL TRIAL: NCT01740102
Title: Does Remote Ischemic Preconditioning Reduce the Incidence of Postoperative Atrial Fibrillation in Patient Undergoing Coronary Artery Bypass Graft Surgery?
Brief Title: Clinical Value of Remote Ischemic Preconditioning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Helse Nord-Trøndelag HF (Other); Namsos Hospital (Other); Sykehuset Innlandet HF (Other); Helse Møre og Romsdal HF (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2011/2525
Record Dates: First submitted 2012-11-21; First posted 2012-12-04 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Heart Diseases; Atrial Fibrillation
Keywords: Ischemic preconditioning; Coronary artery bypass; Preoperative care; Postoperative period
MeSH Terms: conditions — Heart Diseases; Atrial Fibrillation | interventions — Ischemic Preconditioning

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- RIPC (Experimental): Remote ischemic preconditioning (RIPC) in the operating theatre after induction of anaesthesia and before surgery.
  Interventions: Procedure: RIPC
- No RIPC (No Intervention): Patients in the control group will not receive remote ischemic preconditioning before the surgery.

INTERVENTIONS:
Procedure: RIPC — The remote ischemic preconditioning will consist of three sequential sphygmomanometer cuff inflations. The cuff will be inflated up to 200 mmHg for 5 minutes and then deflated for 5 minutes. This cycle will be performed three times in total. The entire preconditioning will therefore last for 25 minutes.
  Other Names: Remote ischemic preconditioning; Ischemic preconditioning
  Arms: RIPC

SUMMARY:
Objectives: Despite utilization of available means for cardioprotection during cardiac surgery, myocardial injury still occurs. Further improvement of cardioprotection is therefore necessary. Remote ischemic preconditioning (RIPC) is an easy and non-invasive method. Laboratory research has shown promising results regarding myocardial survival during open heart surgery, but the clinical value of RIPC is still largely unknown. The investigators hypothesize that RIPC before coronary artery bypass grafting (CABG) reduces the incidence of postoperative atrial fibrillation (POAF).

ELIGIBILITY:
Inclusion Criteria:

* Elective isolated on-pump CABG surgery
* Informed consent

Exclusion Criteria:

* Patients with a severe pulmonary disease
* Patients with renal failure (GFR<30 mL/min/1.73 m2)
* Patients with liver failure
* Peripheral vascular disease affecting the upper limbs
* Patients on sulfonylurea derivatives.
* Patients with atrial fibrillation in their case history
* Prior cardiac surgery (Re-operations)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2012-08; Primary Completion 2013-01 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Postoperative atrial fibrillation | Up to 10 days after surgery
  A patient will be classified as belonging to the postoperative atrial fibrillation group if they have any episode of atrial fibrillation, measured by telemetry, lasting more than 1 minute during their postoperative days at the hospital.

SECONDARY OUTCOMES:
Length of hospital stay | Maximum 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Wahba, MD prof, Study Director — Faculty of Medicine Norwegian University of Science and Technology Trondheim, Norway, and Department of Cardiothoracic Surgery, St. Olavs Hospital, Trondheim, Norway.; Lars Erik B Krogstad, Principal Investigator — Faculty of Medicine Norwegian University of Science and Technology Trondheim, Norway.
Locations (1):
- St Olavs Hospital Trondheim University Hospital, Trondheim, Norway

REFERENCES:
- [Result] Krogstad LE, Slagsvold KH, Wahba A. Remote ischemic preconditioning and incidence of postoperative atrial fibrillation. Scand Cardiovasc J. 2015 Jun;49(3):117-22. doi: 10.3109/14017431.2015.1010565. Epub 2015 Feb 24. PMID 25613907